CLINICAL TRIAL: NCT07248436
Title: "Investigation of the Validity and Reliability of the Pelvic Floor Distress Inventory-20 in Individuals With Primary Sjögren's Syndrome."
Brief Title: "Validity and Reliability of Pelvic Floor Distress Inventory-20 in Primary Sjögren's Syndrome"
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Begüm AKAR, Principal investigator, Pamukkale University
Other Study IDs: Pamukkale U
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Sjogren Syndrome
Keywords: Sjogren syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sjogren syndrome: The Sjogren syndrome group will consist of patients over the age of 18 who apply to the Rheumatology Department of Pamukkale University and meet the inclusion criteria.
  Interventions: Other: the validity and reliability study

INTERVENTIONS:
Other: the validity and reliability study — "To obtain the validity and reliability of the questionnaire in individuals with Sjögren's syndrome."

SUMMARY:
The aim of this study is to examine the Turkish validity and reliability of the Pelvic Floor Distress Inventory-20 in patients with pSS.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Primary Sjögren's Syndrome by the PAÜ Rheumatology clinic
* Being between the ages of 18 and 65
* Volunteering to participate in the study

Exclusion Criteria:

* Presence of neurological disease
* Presence of any orthopedic problem that may affect functionality
* History of orthopedic surgery
* Presence of psychiatric disorder that may affect cooperation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Sjogren syndrome group
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  The patient is asked to rate their complaints of fatigue, pain, and dryness on a scale from 1 to 10, and the arithmetic average of the scores obtained from these three questions is calculated. An ESSPRI score below 5 is considered an acceptable disease status, while a score of 5 or above is considered an indicator of high disease activity.
Pelvic Floor Distress Inventory-20 (PTDE-20) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  There are 20 questions in total on the scale. The best score that can be obtained from the entire survey is "0" and the worst score is "300".
Visual Analog Scale (VAS) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  VAS is used to convert certain values that cannot be measured numerically into numerical form. The patient is asked to indicate where their condition fits on this line by drawing a line, placing a dot, or marking a point. It is evaluated on a scale from 0 to 10.

SECONDARY OUTCOMES:
Cognitive Exercise Therapy Approach (BETY) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  This scale has 30 items. The scale is scored with a 5-point Likert system.
Health assessment questionnaire (HAQ) | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  This questionnaire consists of 20 questions and 8 subheadings, each answer ranging from 0 to 3 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale Üniversitesi, Pamukkale, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No